CLINICAL TRIAL: NCT07386080
Title: The Safety of Carbergoline Versus Placebo for Antipsychotic Induced Hyperprolactinemia: A Pragmatic, Randomised, Non-inferiority Trial With Blinded Outcome.
Brief Title: Carbergoline for Antipsychotic Induced Hyperprolactinemia.
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Zealand University Hospital (Other)
Collaborators: Region Zealand (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: JK-1002
Record Dates: First submitted 2026-01-27; First posted 2026-02-04 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-01

CONDITIONS: Scizophrenia
Keywords: prolactin; cabergoline
MeSH Terms: interventions — Cabergoline; Dopamine Agonists

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Placebo (Placebo Comparator): Placebo tablets + standard care
  Interventions: Drug: Placebo
- Intervention (Active Comparator): Cabergoline tablets + standard care
  Interventions: Drug: Cabergoline (Dopamine Agonist)

INTERVENTIONS:
Drug: Cabergoline (Dopamine Agonist) — This intervention will use cabergoline for antipsychotic induced hyperprolactinemia.
  Arms: Intervention
Drug: Placebo — Placebo + standard care
  Arms: Placebo

SUMMARY:
The goal of this clinical trial is to learn if cabergoline is safe to use in patients with antipsychotic-induced hyperprolactinemia in adults with scizophrenia. The main question it aims to answer :

Is the severity of positive and negative symptoms affected by the use of cabergoline?

Researchers will compare cabergolin to placebo to see if positive and negative symptoms are equel in both groups.

Participants will, in a blinded manor, take either placebo tablets or cabergoline for 12 weeks. The severity of positive and negative symptoms will be evaluated before and after the intervention in both groups.

DETAILED DESCRIPTION:
Antipsychotic (AP) medication is the cornerstone of treatment in patients with schizophrenia, but may be used in patients with depression, severe anxiety, or bipolar disorders. The main regulator of prolactin is exerted by the inhibitory effect of hypothalamic dopamine through its agonistic effects on pituitary D2-receptors. The majority of antipsychotic drugs require a 50 to 60% antagonistic occupancy of the D2 receptor for optimal effect, which explains why hyperprolactinemia is observed in 30% to 70% of patients on AP treatment. Hyperprolactinemia may cause gynecomastia, galactorrhea, infertility, menstrual irregularities, osteopenia, sexual dysfunction, and erectile dysfunction in men, while metabolic and cardiovascular disturbances are currently debated5 - serious side effects that may contribute to the low adherence rates of antipsychotic treatment in patients with schizophrenia spectrum disorders. The consistent association between lack of adherence to treatment and hospitalisation, acute care utilization, and relapse prevention highlights the importance of safe antipsychotic treatment with acceptable side effects. Unacceptable side effects to AP treatment may incline patients and physicians to abandon otherwise successful AP treatment and pursue treatment with less potent antipsychotic properties but with fewer and acceptable side effects. Since 2015, the proportion of Danish citizens treated with antipsychotics has increased every year up to 144.000 in 2023, corresponding to an increase of 19% in less than a decade.

While the effect of prolactin on breast tissue is a direct result of prolactin binding to prolactin receptors the other symptoms of hyperprolactinemia are mainly indirect through reduced gonadotropin levels, i.e. estrogen and testosterone; high prolactin levels result in decreased kisspeptin in the hypothalamus and consequently gonadotropin-releasing hormone (GnRH) release is reduced which leads to lower secretion of luteinizing hormone (LH) and follicle-stimulating hormone (FSH), which is then followed by lower levels of estradiol and testosterone. It could also be hypothesised that hyperprolactinemia may have unwarranted metabolic effects, as often observed in patients in antipsychotic treatment. Current strategies for reducing antipsychotic induced hyperprolactinemia include a change of AP treatment, aripiprazole, estrogen or testosterone supplementation, metformin, or a dopamine receptor agonist (DRA) - i.e. cabergoline or bromocriptine. Once effective APT has been established, changing or reducing the drug or dose is often not desirable, and only aripiprazole, metformin, and DRAs will address both direct and indirect effects of hyperprolactinemia. From an endocrine perspective, treatment with DRAs is tempting due to the fast and highly effective prolactin-lowering properties, the low prevalence of side effects, and administration once or twice weekly (cabergoline).

However, from a theoretical point DRA-treatment may be problematic due to the opposing effects of antipsychotics and DRAs on the dopamine receptor, which may cause exacerbations of psychotic symptoms, which is why endocrinologists are reluctant to introduce DRAs for AP-induced hyperprolactinemia. However, several observational studies have shown significant effect of DRAs on prolactin levels and symptoms associated with AP induced hyperprolactinemia without any adverse effects to psychopathological status, while one RCT found worsening of psychotic symptoms in 1/2018 comparing bromocriptine with a herbal product and only one RCT has examined bromocriptine versus placebo in 60 patients without identifying any worsening in psychopathology. None of the RCT's used blinded outcome assessment, and none of the studies used cabergoline, which is the dopamine receptor agonist with the least number of adverse events, and only requires administration once or twice weekly.

Main objective • Assessing the safety of cabergoline for antipsychotic induced hyperprolactinemia in men and pre-menopausal women with schizophrenia spectrum disorders concerning positive and negative symptoms in a randomised, parallel group, non-inferiority trial with blinded outcome assessment.

Main hypothesis

• We hypothesise that the severity of positive and negative symptoms in participants with antipsychotic induced hyperprolactinemia receiving cabergoline is non-inferior to placebo after 12 weeks of intervention.

Perspective With the high prevalence of AP-induced hyperprolactinemia, the use of cabergoline for augmentation of both direct and indirect effects of high prolactin levels would offer patients an effective prolactin-lowering strategy, few side effects, and allow patients to stay on effective antipsychotic treatment. With a convincing and safe treatment for AP-induced hyperprolactinemia, we expect a larger proportion of patients to be able to remain on the best AP-treatment with no or reduced side-effects from hyperprolactinemia. With the addition of clear guidelines, the treating psychiatrist may, in the future, treat AP-induced hyperprolactinemia themselves rather than referring to an endocrinologist and risk treatment delay. Reducing prolactin levels with cabergoline may also contribute to an improved metabolic profile as observed in patients with type 2 diabetes or hyperprolactinemia.

Method Design: A pragmatic randomised controlled parallel group non-inferiority study with blinded outcome assessment.

ELIGIBILITY:
Inclusion Criteria:

* receiveing antipsychotic treatment for at least 3 months for a schizophrenia spectrum disorder
* Prolactin levels > URL
* symptoms of hyperprolactinemia according to he UKU side effect scale (Udvalg for Klinisk Undersøgelser)
* no suicide ideation at time of recruitment (≤ 2 Columbia-Suicide Serverity Rating Scale)

Exclusion Criteria:

* patients that has previously responded unfavorably to treatment with a dopamine receptor agonist.
* The use of recreational drugs that may give hyperprolactinemia.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — The study only accepts participants with in which biological sex and gender identity is aligned. This is partly due to the studies ability to identify side effects of high prolactin levels, i.e. lack of periods, breast discharge and partly due to biochemical assessment of gonadotropines and prolactin which is specific to the biological sex.
Enrollment: 146 (Estimated)
Dates: Start 2026-05-01 (Estimated); Primary Completion 2028-05-01 (Estimated); Study Completion 2029-05-01 (Estimated)

PRIMARY OUTCOMES:
Total score on the PANSS (Positive and Negative Syndrome Scale) | At end of intervention, i.e. 12 weeks from baseline.
  The primary outcome is the total score of the PANSS in absolute numbers at the end of intervention (12 weeks) comparing the placebo group with the intervention group (cabergoline).

CONTACTS AND LOCATIONS:
Overall Officials: Jesper Krogh, Principal Investigator — Zealand University Hospital
Locations (1):
- Zealand University Hospital, Køge, Region Sjælland, Denmark

IPD SHARING:
Plan to Share IPD: Undecided
IPD data will be shared upon reasonable request provided that a data sharing agreement can bee reached and that the local ethical committee will accept.

REFERENCES:
- [Background] Kuroki T, Watanabe Y, Yamai S, Obara Y, Takizawa K. [Detection of Neisseria gonorrhoeae antigens by an enzyme immunoassay (Gonozyme)]. Kansenshogaku Zasshi. 1985 Dec;59(12):1236-40. doi: 10.11150/kansenshogakuzasshi1970.59.1236. No abstract available. Japanese. PMID 3938800
- [Background] Gonzalez-Rodriguez A, Labad J, Seeman MV. Antipsychotic-induced Hyperprolactinemia in aging populations: Prevalence, implications, prevention and management. Prog Neuropsychopharmacol Biol Psychiatry. 2020 Jul 13;101:109941. doi: 10.1016/j.pnpbp.2020.109941. Epub 2020 Mar 31. PMID 32243999
- [Background] Lang K, Meyers JL, Korn JR, Lee S, Sikirica M, Crivera C, Dirani R, Menzin J. Medication adherence and hospitalization among patients with schizophrenia treated with antipsychotics. Psychiatr Serv. 2010 Dec;61(12):1239-47. doi: 10.1176/ps.2010.61.12.1239. PMID 21123409